CLINICAL TRIAL: NCT06538675
Title: Process and Outcome Evaluation of Psychotherapeutic Approaches At the Outpatient Clinic for Psychotherapy of the Paris Lodron University Salzburg
Brief Title: Process and Outcome Evaluation of Different Psychotherapies
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Salzburg (Other)
Responsible Party: Principal Investigator, Thomas Probst, Professor for Psychotherapy and Psychotherapy Research (Paris Lodron University Salzburg), University of Salzburg
Other Study IDs: 14/2024
Record Dates: First submitted 2024-07-15; First posted 2024-08-06 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-08

CONDITIONS: Mental Illness; Psychiatric Disorder; Mental Disorder
Keywords: psychotherapy
MeSH Terms: conditions — Mental Disorders | interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- psychoanalytic-psychodynamic therapy
  Interventions: Other: Psychotherapy
- humanistic therapy
  Interventions: Other: Psychotherapy
- systemic therapy
  Interventions: Other: Psychotherapy
- cognitive-behavioral therapy
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy — Patients are assigned to a therapist and will receive psychotherapy

SUMMARY:
In this study, adult patients and therapists at the Outpatient Clinic for Psychotherapy of the Paris Lodron University Salzburg will complete questionnaires throughout the course of psychotherapy in order to evaluate the course and outcome of psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients: indication for psychotherapy, adult patients capable of giving consent, with sufficient knowledge of German to complete the questionnaires, signed treatment contract and declaration of consent
* Psychotherapists: officially registered psychotherapists and psychotherapists in training under supervision (in Austria), signed work contract and declaration of consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals seeking help for their mental health at Outpatient Clinic for Psychotherapy of the Paris Lodron University Salzburg.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist Short Form (HSCL-11) | through study completion, an average of 1 year
  11 items, Likert scale: 4-point scale; 1 (not at all) to 4 (very much), Minimum value: 11, Maximum value: 44, Higher scores indicate more mental health problems.

SECONDARY OUTCOMES:
Patient Health Questionnaire-8 (PHQ-8) | through study completion, an average of 1 year
  8 items, Likert scale: 4-point; 0 (not at all) to 3 (nearly every day), Minimun value: 0, Maximum value: 24, Higher scores indicate more depressive symptoms, Score ≥ 10 indicate depression.
Generalizied Anxiety Disorder Scale-7 (GAD-7) | through study completion, an average of 1 year
  7 items, Likert scale: 4-point; 0 (not at all) to 3 (nearly every day), Minimun value: 0, Maximum value: 21, Higher scores indicate more anxiety symptoms, Score ≥ 10 indicate anxiety.
Patient Health Questionnaire-4 (PHQ-4) | through study completion, an average of 1 year
  4 items, Likert scale: 4-point; 0 (not at all) to 3 (nearly every day), Minimun value: 0, Maximum value: 12, Higher scores indicate more depressive and anxiety symptoms, Score ≥3 for first 2 questions indicates depression, Score ≥ 3 for last 2 questions indicates anxiety.
Positive Mental Health scale (PMH) | through study completion, an average of 1 year
  9 items, Likert skala: 4-point; 0 (do not agree) to 3 (agree), Minimun value: 0, Maximum value: 27, Higher scores indicate higher positive mental health.
Society for Psychotherapy Research Item on Mental Health | through study completion, an average of 1 year
  1 item, Likert scale: 5-point; 0 (very bad) to 4 (very good), Minimum value: 0, Maximum value: 4, Higher scores indicate better mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Probst, Univ.Prof.Dr, Study Director — Paris-Lodron-University Salzburg; Franziska Pfannerstill, Dr., Principal Investigator — Paris-Lodron-University Salzburg; Hannah van Alebeek, Dr., Principal Investigator — Paris-Lodron-University Salzburg
Locations (1):
- Paris-Lodron-University Salzburg, Salzburg, Salzburg, Austria

REFERENCES:
- See also: Related Info — http://www.plus.ac.at/psychotherapie